CLINICAL TRIAL: NCT04477642
Title: Abatacept for Patients With COVID-19 and Respiratory Distress
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Children's Hospital (Other); Bristol-Myers Squibb (Industry); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-P-00XXX
Record Dates: First submitted 2020-04-22; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AbataceptTreatment Arm (Experimental): Enrolled patients who will receive treatment with abatacept
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — 10mg/kg intravenously administered on Day 1

SUMMARY:
This is a single-arm open label trial for hospitalized patients with COVID-19 (Coronavirus). The primary endpoint of the study is to assess the requirement for mechanical ventilation in patients who are admitted to the hospital with COVID-19 infection and a Pulse Oxygen Level </= 93% on room air. The primary endpoint analysis will be performed using all enrolled patients.

DETAILED DESCRIPTION:
Patients with COVID-19 who are admitted with respiratory distress will be considered for enrollment on this study. Patients will be screened and then if they meet eligibility criteria will be enrolled. Abatacept will be administered on Day 1 at a dose of 10 mg/kg. Patients will then be followed closely through 90 days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Confirmed SARS-CoV-2 infection, confirmed by polymerase chain reaction (PCR) </=4 days prior to enrollment
* Evidence of respiratory distress including SpO2 </=93% on room air.
* Radiographic evidence of pulmonary infiltrates.
* Ability to understand and the willingness to provide informed consent.

Exclusion Criteria:

* Patients already intubated/mechanically ventilated at screening will not be eligible.
* Patients with uncontrolled severe bacterial or fungal infections at the time of enrollment.
* Patients with previously diagnosed autoimmune disorders or who were on immunosuppressive medications prior to developing COVID-19 are not eligible
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation-free survival | 30 days
  Cumulative incidence of mechanical ventilation-free survival at 30 days after initiation of abatacept

SECONDARY OUTCOMES:
Duration of days on a ventilator | 30 days
  Number of days a patient is on a ventilator, if applicable
Days until pulse oxygen is > 93% on room air | 30 days
  Number of days until patient recovers with SpO2 > 93%
Days until supplemental oxygen is no longer required | 30 days
  No supplemental oxygen for at least 24 hours
Duration of fever >= 38°C | 30 days
  Number of days until fever is less than 38°C
Overall survival | 90 days
  Patient survival status through 90 days
Infusion reactions | 14 days
  Number of Infusion Reactions in patients treated with abatacept
Secondary infections | 90 days
  Number of Secondary infections in patients treated with abatacept
Change in Clinical Status, based on 7-point ordinal scale | 14 days
  Change in clinical status from baseline, as assessed by a 7-point ordinal scale on Day 14
Viral load | 28 days
  Viral load at baseline and on Days 7, 14, 21, 28 (each +/- 2 days) after the first abatacept dose.
Radiographic Improvement | 14 days
  Improvement in lung findings based on CXR (chest x-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts